CLINICAL TRIAL: NCT02515097
Title: A Phase 3, Multicenter, Double-Blind, Randomized, Vehicle Controlled Clinical Study to Assess the Safety and Efficacy of IDP-122 in the Treatment of Plaque Psoriasis
Brief Title: Safety and Efficacy of IDP-122 in the Treatment of Participants With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-122A-302
Record Dates: First submitted 2015-07-31; First posted 2015-08-04 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-122 Lotion (Experimental): Participants will apply IDP-122 Lotion (halobetasol propionate [HP] 0.01%) topically once daily for 8 weeks.
  Interventions: Drug: IDP-122 Lotion
- IDP-122 Vehicle Lotion (Placebo Comparator): Participants will apply IDP-122 Vehicle Lotion topically once daily for 8 weeks.
  Interventions: Drug: IDP-122 Vehicle Lotion

INTERVENTIONS:
Drug: IDP-122 Lotion — Medicated topical lotion
  Other Names: HP 0.01%
  Arms: IDP-122 Lotion
Drug: IDP-122 Vehicle Lotion — Vehicle topical lotion with no active ingredient
  Arms: IDP-122 Vehicle Lotion

SUMMARY:
This study is to evaluate the safety and efficacy of a topical lotion when applied once daily to adult participants with moderate to severe plaque psoriasis (defined as an Investigator's Global Assessment [IGA] score of 3 or 4).

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and efficacy of topical IDP-122 Lotion when applied once daily to adult participants with moderate to severe plaque psoriasis. The intent of the study is specifically to evaluate the safety and efficacy of a once daily application of IDP-122 Lotion in comparison with vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a body surface area (BSA) of at least 3%, but no more than 12%. The face, scalp, palms, soles, axillae, and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an IGA score of 3 or 4. (The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this assessment).

Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the Investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the Investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the Investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half-lives (whichever is longer) prior to the Baseline visit or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, Study Director — Valeant Pharmaceuticals
Locations (15):
- United States (15):
  - Valeant Site 14, Santa Ana, California
  - Valeant Site 02, Boynton Beach, Florida
  - Valeant Site 10, Clearwater, Florida
  - Valeant Site 1, Tampa, Florida
  - Valeant Site 07, Plainfield, Indiana
  - Valeant Site 15, Olathe, Kansas
  - Valeant Site 08, Fridley, Minnesota
  - Valeant Site 13, Omaha, Nebraska
  - Valeant Site 04, New York, New York
  - Valeant Site 12, Stony Brook, New York
  - Valeant Site 05, High Point, North Carolina
  - Valeant Site 11, Knoxville, Tennessee
  - Valeant Site 03, Houston, Texas
  - Valeant Site 09, San Antonio, Texas
  - Valeant Site 06, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- IDP-122 Lotion: Participants applied IDP-122 Lotion (halobetasol propionate [HP] 0.01%) topically once daily for 8 weeks.
- IDP-122 Vehicle Lotion: Participants applied IDP-122 Vehicle Lotion topically once daily for 8 weeks.
Period: Overall Study
Arm/Group | IDP-122 Lotion | IDP-122 Vehicle Lotion
Started | 142 | 71
Intent-to-Treat (ITT) Population (Participants who were randomized and dispensed study drug.) | 142 | 71
Safety Population (Randomized participants with ≥1 confirmed dose of study drug and ≥1 post-Baseline safety assessment.) | 142 | 70
Completed | 135 | 65
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and dispensed study drug (ITT population).
Groups:
- IDP-122 Lotion: Participants applied IDP-122 Lotion (HP 0.01%) topically once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | IDP-122 Lotion | IDP-122 Vehicle Lotion | Total
Number analyzed (Participants) | 142 | 71 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.31) | 53.4 (12.73) | 53.9 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 29 | 84
  Male | 87 | 42 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 23 | 58
  Not Hispanic or Latino | 107 | 48 | 155
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4 | 2 | 6
  Black or African American | 12 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 122 | 61 | 183
  Mexican | 0 | 1 | 1
  Puerto Rican | 0 | 1 | 1
  South Asian | 0 | 1 | 1
  Philipino | 0 | 1 | 1
  Mixed | 1 | 1 | 2
  Unknown | 3 | 0 | 3
Investigator's Global Assessment [IGA] Score [Number; unit: participants] — The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe).
  participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 0 | 0 | 0
    3 - Moderate | 124 | 65 | 189
    4 - Severe | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Success at Week 8
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the IGA score and an IGA score equating to "clear" or "almost clear" at Week 8. The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe). The face, scalp, palms, soles, axillae, and intertriginous areas were excluded from this assessment.
Time Frame: Week 8
Population: Participants who were randomized and dispensed study drug (ITT population). Markov Chain Monte Carlo (MCMC) multiple imputation was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | IDP-122 Lotion | IDP-122 Vehicle Lotion
Number analyzed (Participants) | 142 | 71
percentage of participants | 38.41 | 11.99

2. Secondary Outcome: Percentage of Participants With Treatment Success at Weeks 2, 4, 6, and 12
Description: Treatment success defined as at least a 2-grade improvement from Baseline in the Investigator's Global Assessment (IGA) score and an IGA score equating to "clear" or "almost clear" at Weeks 2, 4, 6, and 12. The IGA score was based on a 5-point scale ranging from 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, and 4=severe). The face, scalp, palms, soles, axillae, and intertriginous areas were excluded from this assessment.
Time Frame: Weeks 2, 4, 6, and 12 (4-week follow-up)
Population: Participants who were randomized and dispensed study drug (ITT population). MCMC multiple imputation was used to impute missing data.
Measure: Number; unit: percentage of participants
Arm/Group | IDP-122 Lotion | IDP-122 Vehicle Lotion
Number analyzed (Participants) | 142 | 71
percentage of participants
  Week 2 | 4.93 | 0.00
  Week 4 | 19.26 | 0.20
  Week 6 | 27.71 | 4.35
  Week 12 | 23.04 | 9.34

ADVERSE EVENTS:
Time Frame: Baseline through Week 12
Description: Adverse events were collected from participants who were randomized, received at least 1 confirmed dose of study drug, and had at least 1 post-Baseline safety assessment (Safety Population).
Arm/Group | IDP-122 Lotion | IDP-122 Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 1/142 | 0/71
Serious Adverse Events (participants affected / at risk) | 2/142 | 1/71
Other Adverse Events (participants affected / at risk) | 0/142 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-122 Lotion (N=142) | IDP-122 Vehicle Lotion (N=71)
Myocardial infarction (Cardiac disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT02515097/Prot_SAP_000.pdf